CLINICAL TRIAL: NCT00360581
Title: Preventing Postpartum Relapse to Smoking Using Yoga and Cognitive Behavioral Therapy: A Randomized Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0603012
Record Dates: First submitted 2006-08-02; First posted 2006-08-04 (Estimated); Last update posted 2008-02-11 (Estimated); Status verified 2008-02

CONDITIONS: Smoking Cessation
Keywords: Smoking abstinence
MeSH Terms: conditions — Smoking Cessation | interventions — Yoga; Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Yoga
Behavioral: Yoga and Cognitive Behavioral Therapy

SUMMARY:
The purpose of this study is to develop strategies to maintain smoking abstinence initiated in pregnancy and prevent relapse in the postpartum period.

DETAILED DESCRIPTION:
Many women quit smoking during pregnancy, but postpartum relapse rates are high, approximately, 50-80% (Van't Hof, et al). The majority of women who quit smoking during pregnancy resume smoking within the first 3 months postpartum (McBride, et al). The environmental risks of tobacco smoke on the newborn child can lead to acute respiratory infections, bronchitis, pneumonia, and SIDS. Several studies have tried to identify reasons for the high rates of relapse. Postpartum relapse has been attributed to decreased self-efficacy, the lack of effective coping strategies to resist temptation to smoke, and weight concerns (McBride, et al). Addictive behaviors such as smoking are learned behavioral means of coping. By learning new rules for dealing with problems, a behavior can be modified or unlearned. Physical exercise, when combined with cognitive behavioral therapy (CBT) as a smoking cessation treatment, is useful in the maintenance of smoking cessation in women. Yoga, as a form of exercise, has been shown to promote the desire to stop smoking and enhance subjective well-being and mood. Though untested in postpartum relapse prevention, yoga practice, when coupled with CBT, may address both mood and physiologic postpartum sensations that may be associated with the prevention of smoking relapse. Women are more apt to decrease or even stop smoking during pregnancy, and if successful in sustaining cessation, are likely to live longer.

This randomized exploratory pilot study will use a controlled parallel group design using smoking cessation yoga intervention and cognitive behavioral therapy. The study will include a total of 30 participants aged 18-45 years. Smoking status will be identified by self-report and carbon monoxide testing at enrollment. At randomization and following time points, smoking status will be identified by self-report and confirmed by carbon monoxide testing.

ELIGIBILITY:
Inclusion Criteria:

* Must have the ability to read, write, and understand English.
* Must have quit smoking during their current pregnancy.
* Must possess the desire to remain smoke-free after delivery.
* Obtain permission from obstetrician to participate in yoga.
* Must be reachable by telephone.
* If subject becomes pregnant again while in the study, she can still participate with written permission from her primary care physician.

Exclusion Criteria:

* Untreated hypertension.
* A history of: glaucoma, major depression, alcohol abuse or substance disorder, anorexia nervosa, or head trauma.
* Recent abdominal surgery (such as caesarean section).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-04; Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
smoking abstinence by CO testing

SECONDARY OUTCOMES:
smoking abstinence by self-report

CONTACTS AND LOCATIONS:
Overall Officials: Susan A. Albrecht PhD, RN, FAAN, Principal Investigator — University of Pittsburgh School of Nursing
Locations (1):
- University of Pittsburgh School of Nursing, Pittsburgh, Pennsylvania, United States